CLINICAL TRIAL: NCT04980625
Title: Safety and Efficacy of Remote Ischemic Conditioning Combined With Intravenous Thrombolysis for Acute Ischemic Stroke: A Multicenter, Randomized, Parallel-controlled Clinical Trial
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning Combined With Intravenous Thrombolysis for Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERIC-IVT
Record Dates: First submitted 2021-07-13; First posted 2021-07-28 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+Standard medical treatment (Active Comparator): RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 consecutive days from thrombolysis. Additionally, the patients will be treated with standard medical treatment according to the Guidelines for diagnosis and treatment of acute ischemic stroke in China.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+Standard medical treatment (Placebo Comparator): Sham RIC+Standard medical treatment Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 consecutive days from thrombolysis. Additionally, the patients will be treated with standard medical treatment according to the Guidelines for diagnosis and treatment of acute ischemic stroke in China.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mm Hg.
  Arms: RIC+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Sham remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mm Hg.
  Arms: Sham RIC+Standard medical treatment

SUMMARY:
The purpose of this study is to determine the efficacy and safety of remote ischemic conditioning combined with intravenous thrombolysis in treating acute ischemic stroke.

DETAILED DESCRIPTION:
In this study, 558 cases of ischemic stroke who undergo intravenous thrombolysis within 4.5 hours from the onset are included in 18 centers in China according to the principle of random, and parallel control. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 7 consecutive days. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day for 7 consecutive days. Two groups will be followed up for 90 days to evaluate the efficacy and safety of remote ischemic conditioning combined with intravenous thrombolysis in treating acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age≥18 years, regardless of sex;
* 2) Patients with a clinically definite diagnosis of acute ischemic stroke and undergo intravenous thrombolysis with alteplase;
* 3) Pre-thrombolysis NIHSS >= 4, and <= 24;
* 4) Premorbid mRS 0-1;
* 5) Signed and dated informed consent is obtained;

Exclusion Criteria:

* 1) Patients who have the contraindication of intravenous thrombolysis with alteplase.
* 2) The patients who have the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb.
* 3) Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc.
* 4) Pregnant or lactating women.
* 5) Severe hepatic and renal dysfunction.
* 6) Patients with a life expectancy of less than 3 months or patients unable to complete the study for other reasons.
* 7) Unwilling to be followed up or treated for poor compliance.
* 8) He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission.
* 9) Other conditions that the researchers think are not suitable for the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Modified Rankin Scale (mRS) Score 0-1 | 3 months
  Proportion of patients with Modified Rankin Scale (mRS) Score 0-1. Ranged from 0 to 6, a low value represents a better outcome.

SECONDARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) at 24 hours, and 7 days after IVT. | 24 hours, 7 days
  National Institute of Health stroke scale (NIHSS) at 24 hours, and 7 days after IVT. Ranged from 0 to 42, a low value represents a better outcome.
Barthel Index (BI) at 24 hours, and 7 days after IVT. | 24 hours, 7 days
  Barthel Index (BI) at 24 hours, and 7 days after IVT. Ranged from 0 to 100, a high value represents a better outcome.
Proportion of patients with modified Rankin Scale (mRS) Score 0-2 at 90±3 days after IVT. | 90±3 days
  Proportion of patients with modified Rankin Scale (mRS) Score 0-2 at 90±3 days after IVT. mRS: Ranged from 0 to 6, a low value represents a better outcome.
Frequency of adverse events during follow-up | 90 days
  All adverse events through 90 days.
Frequency of Hemorrhagic transformation within 24 hours after IVT. | 24 hours
  Frequency of Hemorrhagic transformation within 24 hours after IVT.
Mortality within 90 days. | 90 days
  Mortality within 90 days.
Stroke recurrence rate within 90 days. | 90 days
  Stroke recurrence rate within 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Guo ZN, Abuduxukuer R, Zhang P, Qu Y, Wang LJ, Zhao JF, Ju DS, Wang JM, Jin HM, Wang WW, Teng RH, Gao JH, Yuan ZM, Gao HF, Jiang YF, Li ZD, He Y, Jiang LG, Li L, Hu XF, Jiang CL, Wang R, Qi YB, Xin H, Jia Y, Yu H, Jin H, Chen HS, Wang DL, Nguyen TN, Yang Y; SERIC-IVT study group. Safety and Efficacy of Remote Ischemic Conditioning in Patients With Intravenous Thrombolysis: The SERIC-IVT Trial. Stroke. 2025 Feb;56(2):335-343. doi: 10.1161/STROKEAHA.124.048509. Epub 2025 Jan 8. PMID 39772709